CLINICAL TRIAL: NCT03826641
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1801 in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1801 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-DAME-101
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1 : Fasted state + HCP1805, Period 2 : Fasted state + HCP1801
  Interventions: Drug: HCP1805; Drug: HCP1801
- Sequence 2 (Experimental): Period 1 : Fasted state + HCP1801, Period 2 : Fasted state + HCP1805
  Interventions: Drug: HCP1805; Drug: HCP1801
- Sequence 3 (Experimental): Period 1 : High fat diet + HCP1805, Period 2 : High fat diet + HCP1801
  Interventions: Drug: HCP1805; Drug: HCP1801
- Sequence 4 (Experimental): Period 1 : High fat diet + HCP1801, Period 2 : High fat diet + HCP1805
  Interventions: Drug: HCP1805; Drug: HCP1801

INTERVENTIONS:
Drug: HCP1805 — Dapagliflozin/Metformin (Xigduo XR) 10/1000mg
Drug: HCP1801 — Dapagliflozin/Metformin 10/1000mg

SUMMARY:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics, safety and tolerability of HCP1801 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Cmax of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
AUClast of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Cmax of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
AUClast of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Tmax of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
t1/2 of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
CL/F of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Vd/F of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
AUCinf of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Tmax of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
t1/2 of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
CL/F of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Vd/F of Metformin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No